CLINICAL TRIAL: NCT07161440
Title: Steroid Profiling in Adolescents and Young Women With PCOS: Effects of Oral Contraceptive Therapy Assessed by LC-MS/MS
Brief Title: Steroid Profiles in PCOS and Effect of OCP Treatment
Acronym: PCOSLCMS
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Ozge Bayrak Demirel, Pediatric Endocrinologist, Istanbul University
Other Study IDs: PEDENDO-ITF-PCOS-LCMS
Record Dates: First submitted 2025-08-30; First posted 2025-09-08 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Polycystic Ovary Syndrome (PCOS)
Keywords: PCOS; Steroid Profiling; Oral Contraceptives; LC-MS/MS; Adolescents; Hyperandrogenism
MeSH Terms: conditions — Polycystic Ovary Syndrome; Hyperandrogenism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum samples were retained for analysis. These samples were used to assess the steroid profile via liquid chromatography-mass spectrometry (LC-MS/MS). Specifically, levels of intermediate steroid metabolites such as 17-hydroxyprogesterone, androstenedione, testosterone, dehydroepiandrosterone (DHEA), dehydroepiandrosterone sulfate (DHEAS), 11-deoxycortisol, and cortisol were evaluated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PCOS patients without treatment: This cohort included adolescent patients diagnosed with polycystic ovary syndrome (PCOS) who did not receive any medical treatment during the study period. Steroid hormone levels were measured using LC-MS/MS at baseline for all participants to evaluate the endogenous steroid profile in untreated PCOS.
- PCOS patients treated with OCP: This cohort consisted of adolescent patients with polycystic ovary syndrome (PCOS) who were prescribed oral contraceptive pills (OCP) due to clinical indications. A total of 15 patients from the untreated PCOS group received OCP treatment and were followed for 6 months. Baseline and 6-month serum samples were analyzed using liquid chromatography-tandem mass spectrometry (LC-MS/MS) to evaluate changes in steroid hormone profiles after treatment.

SUMMARY:
This prospective observational study investigates the changes in serum steroid intermediates assessed by liquid chromatography-mass spectrometry (LC-MS/MS) in adolescents and young women with polycystic ovary syndrome (PCOS), before and after oral contraceptive (OCP) treatment.

DETAILED DESCRIPTION:
The study enrolled 56 female patients aged 13-21 years with a diagnosis of PCOS according to Rotterdam criteria. At baseline, all participants underwent LC-MS/MS steroid profiling. A subgroup of 15 patients received oral contraceptive therapy based on clinical indication, independent of the study protocol. A second LC-MS/MS steroid analysis was performed at 6 months in this subgroup. The primary aim was to investigate the effect of OCP on the steroid biosynthesis profile. The study was approved by the Istanbul University Ethics Committee (Approval ID: 2019/822) and conducted between January 2020 and December 2021.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PCOS based on Rotterdam criteria
* Age between 13 and 21 years
* No hormonal treatment in the 3 months prior to study enrollment
* Consent provided

Exclusion Criteria:

* Congenital adrenal hyperplasia
* Cushing's syndrome
* Pregnancy
* Use of hormonal medications within 1 year prior to baseline

Ages: 13 Years to 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Adolescent females aged 13 to 21 years diagnosed with polycystic ovary syndrome (PCOS) according to the Rotterdam criteria. All participants were evaluated at the Istanbul Faculty of Medicine between 2020 and 2021. Baseline serum steroid profiles were analyzed using LC-MS/MS in all participants. A subset of 15 patients received oral contraceptive treatment for medical indications and had follow-up hormonal evaluations at 6 months.
Sampling Method: Non-Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2021-01-02 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2025-08-04 (Actual)

PRIMARY OUTCOMES:
Serum adrogen levels | 6 months
  Change in serum androgen levels (e.g., testosterone, androstenedione, DHEAS) measured by LC-MS/MS between baseline and 6 months in the OCP-treated group.
serum androgen levels | 6 months
  Change in serum androgen levels (e.g., testosterone, androstenedione, DHEAS) measured by LC-MS/MS between baseline and 6 months in the OCP-treated group.

SECONDARY OUTCOMES:
Change in serum steroid hormone levels after 6 months of OCP treatment in adolescents with PCOS | Baseline and 6 months after the initiation of OCP treatment
  Comparison of steroid hormone profiles measured by LC-MS/MS between the baseline and 6-month follow-up in adolescent PCOS patients who were treated with oral contraceptive pills (OCP). This outcome aims to assess the impact of OCP therapy on specific androgenic and progestogenic steroid metabolites.

CONTACTS AND LOCATIONS:
Overall Officials: Melek Yildiz, Associate Professor, Principal Investigator — Istanbul University
Locations (1):
- Istanbul University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No